CLINICAL TRIAL: NCT04436354
Title: The Effect of Trendelenburg Lithotomy Position on Pain and Procedural Time During Vaginoscopic Office Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma ketenci gencer, Principle investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GaziosmanpasaTREHa
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2020-06

CONDITIONS: Uterine Diseases
Keywords: vaginoscopic office hysteroscopy; lithotomy position; trendelenburg lithotomy position; visual pain score; procedural time; Likert scale
MeSH Terms: conditions — Uterine Diseases | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaginoscopic office hysteroscopy in the trendelenburg position (Experimental)
  Interventions: Procedure: vaginoscopic office hysteroscopy
- vaginoscopic office hysteroscopy in lithotomy position (Experimental)
  Interventions: Procedure: vaginoscopic office hysteroscopy

INTERVENTIONS:
Procedure: vaginoscopic office hysteroscopy — comparison of procedural time and pain scores of patients in different gynecologycal positions
  Other Names: positions

SUMMARY:
The present study revealed that the TL position is supposed to be more efficient not only for lowering pain score but also reducing the procedural time. Also, performing hysteroscopy in this position may be easier for doctors than in the lithotomy position.

DETAILED DESCRIPTION:
VOH is a widely used diagnostic method and seems to be getting more into outpatient clinics. Despite its huge contribution to clinical practice, pain during the procedure is an important limiting factor. We aimed to investigate the effect of the trendelenburg lithotomy position to the pain and procedural time.However, there is a scarcity of research on this subject. Therefore, the rationale of the study was to enlighten the gap in the literature regarding the pain score and procedural time during VOH for diagnostic purposes in TL position. In order to gain scientific evidence, a randomized controlled trial was conducted to compare pain score and duration of procedure between the standard lithotomy position and TL position. Also, the convenience for the physician performing the procedure was assessed. To the best of our knowledge, this is the first study in the literature investigating the effect of the position of the patient during the procedure on both time, pain, and the convenience for the physician simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* uterine disorders
* abnormal uterine bleeding
* infertility

Exclusion Criteria:

* pregnancy
* cervical disorders
* pelvic infections

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score for pain | 12 months
  The Visual Pain Scale (VPS) was used to evaluate pain levels with 0 represented pain-free, while 10 described the most severe pain (Ekin et al. 2009; Price et al. 1983). Patients were asked to mark the pain expressing point on the VPS immediately after VOH. The severity of pain is determined by the value of the point (cm) marked by the participant
procedural times | 12 months
  minutes

SECONDARY OUTCOMES:
attitudinal Likert type survey | 12 months
  with a 5-point attitudinal Likert type survey; a psychometric scale commonly used to score responses in a questionnaire. The ease or difficulty of the procedure was categorized as 1-very easy, 2-easy, 3-ineffective, 4-difficult, 5-very difficult, and the physician performing the procedure marked
  the appropriate section for each VOH procedure in the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri University Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes